CLINICAL TRIAL: NCT04637776
Title: Psychosocial Syndemics and Multimorbidity in Patients With Heart Failure - R01 HL151431
Brief Title: Psychosocial Syndemics of Heart Failure
Status: Active, not recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Kenneth Freedland, Professor, Washington University School of Medicine
Other Study IDs: 1R01HL151431 (NIH)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Heart Failure: Patients with heart failure who were discharged within the past month after hospitalization for any reason.
  Interventions: Other: Hospitalization

INTERVENTIONS:
Other: Hospitalization — Hospitalization for any reason

SUMMARY:
Heart failure (HF) is a common and debilitating chronic disease with a poor prognosis. Many patients with HFhave psychiatric problems such as depression and other medical disorders such as lung or kidney disease.This study will examine the effects that these psychiatric and medical disorders have on HF outcomes.

DETAILED DESCRIPTION:
Approximately 6.2 million Americans have heart failure (HF) and the prevalence is increasing rapidly. HF is a common cause of hospitalization and mortality in older adults, and the cost of hospital care for HF is skyrocketing. One reason why HF is so burdensome and costly is that it is often complicated by cardiovascular and noncardiovascular comorbidities, especially in older patients. Psychiatric and medical disorders that are risk factors for incident HF persist after HF has developed, and additional comorbidities accumulate as patients with HF grow older. Thus, HF is embedded within a larger pattern of multimorbidity. Unfortunately, most trials of HF therapies as well as many other studies of HF have excluded patients with complex psychiatric and medical comorbidities or severe cognitive impairment. This has left large gaps in research on the care of older adults with HF. In addition, research on socioeconomic risk factors and health disparities has not been integrated with research on multimorbidity in HF. Heart failure is only one of multiple challenges facing patients with multimorbidity, stressful socioeconomic circumstances, and psychosocial problems, but the fragmentation of research on HF has left us with little understanding of patients with complex psychosocial problems. The purpose of this study is to identify combinations of comorbidities and health disparities may affect HF outcomes and require different mixtures of medical, psychological, and social services to address. It will encompass both psychiatric and medical comorbidities but will emphasize the role of psychiatric comorbidities. Syndemics theory is a useful framework for studying this type of psychosocial and medical complexity. Syndemics, also known as synergistic epidemics, occur when there are adverse interactions between prevalent disorders that concentrate in populations that are vulnerable due to adverse socioeconomic or environmental conditions. The syndemics framework has yielded important insights into a number of other disorders, but it has not been used to study the complex psychosocial problems of patients with HF. To our knowledge, this will be the first study of the syndemics of psychiatric and medical comorbidities in heart failure. The multimorbidity framework is an alternative approach for investigating the effects of multiple comorbidities on health outcomes. The specific aims of the study are: 1) to determine the coprevalence of major psychiatric and medical comorbidities in patients with HF (n=535); 2) to determine whether coprevalent comorbidities have synergistic effects on all-cause readmission and mortality risks, heart failure self-care, and perceived global health; 3) to identify vulnerable subpopulations of patients with HF who have higher coprevalences of syndemic comorbidities compared to less vulnerable subpopulations; 4) to determine the extent to which syndemic comorbidities explain adverse HF outcomes (readmissions and mortality, poor self-care, and poor perceived health) in vulnerable subgroups of patients with HF; and 5) to determine the effects of multimorbidity on readmissions, mortality risk, self-care, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from an inpatient hospitalization within the past month, AND
* had a clinical diagnosis of HF at admission to or discharge from the hospital, AND
* met the European Society of HF diagnostic criteria during the hospital stay.

Exclusion Criteria:

* patient's physician advises against participation in the study, OR
* patient refuses to participate, OR
* patient's legally authorized representative refuses to allow patient to participate, OR
* isolated right HF (cor pulmonale), OR
* reversible HF due to valve disease with impending surgical correction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure who were discharged from a hospital in the St. Louis, Missouri area within the past month.
Sampling Method: Non-Probability Sample
Enrollment: 367 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospital readmissions | 4 years or less, depending upon available follow-up time
  Number of hospital readmissions for HF or for other reasons

SECONDARY OUTCOMES:
HF Self-Care | Baseline
  Self-Care of Heart Failure Index v7.2 questionnaire; score range, 0-100 (higher is better)
Global health | Baseline
  PROMIS Global Health V1.2 questionnaire 8-item short form; score range, 0-100 (higher is better)
Medication management | Baseline
  PROMIS Manage Medications questionnaire 4-item short form; score range, 0-100 (higher is better)
Activities of daily living | Baseline
  PROMIS Manage Daily Activities questionnaire 8-item short form; score range, 0-100 (higher is better)
Perceived stress | Baseline
  Perceived Stress Scale (Cohen et al., 1983); score range, 0-40 (higher is worse)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Freedland, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital at Washington University Medical Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be shared on request after the closure of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The dataset is expected to be finalized in mid- to late-2024.
Access Criteria: Affiliation with a recognized research institution

REFERENCES:
- [Derived] Freedland KE, Steinmeyer BC, Skala JA, Carney RM, Rich MW. Patient-Reported Social Determinants of Health in Patients With Heart Failure. J Am Heart Assoc. 2025 May 20;14(10):e041458. doi: 10.1161/JAHA.124.041458. Epub 2025 May 13. PMID 40357673

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT04637776/SAP_000.pdf